CLINICAL TRIAL: NCT04028947
Title: Prophylactic Infrapatellar Saphenous Neurectomy in Primary Total Knee Arthroplasty: A Double-Blind Randomized Controlled Trial
Brief Title: Prophylactic Infrapatellar Saphenous Neurectomy in Primary Total Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Glenn G. Shi, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-000527
Record Dates: First submitted 2019-03-27; First posted 2019-07-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Knee Pain Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard TKA (No Intervention): Subjects will have the standard procedure.
- TKA with Neurectomy (Active Comparator): Subjects will the nerve excised and protected with soft tissue.
  Interventions: Procedure: Prophylactic Infrapatellar Saphenous Neurectomy in Primary Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Prophylactic Infrapatellar Saphenous Neurectomy in Primary Total Knee Arthroplasty — Prophylactic infrapatellar saphenous nerve neurectomy will be performed at the same time as the TKA.
  Arms: TKA with Neurectomy

SUMMARY:
Researchers are trying to determine if knee pain can be reduced by proactively protecting the free end of the saphenous nerve versus leaving it in the standard position during total knee arthroplasty.

DETAILED DESCRIPTION:
Subjects scheduled for total knee arthroplasty will be randomized to two arms. One arm will have the standard saphenous nerve neurectomy during their surgery. The other arm will have the same neurectomy procedure with the free end of the nerve tucked into soft tissue to protect the nerve ending.

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral total knee arthroplasty candidate

Exclusion Criteria:

* Body Mass Index (BMI) >40
* Inflammatory arthritis
* Unable to follow up visits (long distance from Mayo Clinic)
* Poor compliance risk
* Health condition deemed by physician to preclude patient's ability to participate in the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain after surgery | 6 months
  Self-reported pain using Visual Analog Scale which is scored using a horizontal scale from 0-10cm with 10 being the worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn G Shi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials